CLINICAL TRIAL: NCT03866772
Title: Labor Induction With Double Balloon Device, Oral Misoprostol and Concomitant Use of Both. Multicenter Randomized Controlled Trial- IDOM Trial
Brief Title: Labor Induction With Double Balloon Device, Oral Misoprostol and Concomitant Use of Both
Acronym: IDOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: RECRUTIMENT DIFICULTIES
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Inna.bleicher, principle investigator, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0166-18-BNZ
Record Dates: First submitted 2019-03-03; First posted 2019-03-07 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy Related
Keywords: induction of labor; unfavorable cervix; misoprostol; cytotec; double balloon device; cervical ripening
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- MISOPROSTOL (Active Comparator): * oral misoprostol, 50 microgram, every 4 hours
  * Repeat treatment every 4 hours until active labour begins: regular painful contractions (≥ 3 in 10 min), cervical dilatation ≥ 3 cm
  * maximal number of doses: 6
  * Oxytocin infusion can be initiated 4 hours after the last dose of Misoprostol.
  * Failure of induction will be considered if no cervical change nor uterine contractions have begun during 24 hours of treatment.
  * Electronic fetal monitoring should be performed for 30 min after administration of misoprostol and 60 min after any tachysystole.
  Interventions: Drug: Misoprostol Oral Tablet
- DOUBLE BALLOON (Active Comparator): * Insertion of the DBD as instructed by the manufacturer, removal after 6 hours.
  * Artificial rupture of membranes (AROM) if suitable + IV oxytocin administration
  * If AROM cannot be performed- oxytocin infusion will be initiated at first.
  * If Bishop <3 after DBD removal, clinical evaluation and lag time before considering other methods for ripening is suitable and is up to the physician on call.
  Interventions: Device: double balloon device for cervical ripening
- MISOPROSTOL+DOUBLE BALLOON (Active Comparator)
  Interventions: Drug: Misoprostol Oral Tablet; Device: double balloon device for cervical ripening

INTERVENTIONS:
Drug: Misoprostol Oral Tablet — 50 mcg oral consumption
  Arms: MISOPROSTOL; MISOPROSTOL+DOUBLE BALLOON
Device: double balloon device for cervical ripening — insertion for 6 hours and followed by the above mentioned protocol
  Arms: DOUBLE BALLOON; MISOPROSTOL+DOUBLE BALLOON

SUMMARY:
The aim of this study is to compare the rate of cesarean delivery between 3 methods of labor induction: double balloon device, oral misoprostol and combination of the two.

DETAILED DESCRIPTION:
Induction of labor is a common obstetrical procedure. It accounts for 20% of laboring women worldwide.

In the past, studies showed that cesarean delivery rates (CDR) are higher in women who are induced. These studies were comparing induction to spontaneous labor, which is not the management in practice, and when the comparison was made between induction and expectant management, the conclusion was that the induction does not increase CDR and can even reduce its' rate.

Failure of induction depends on the definition, and even among randomized controlled trials, this definition may vary greatly.

The decision whether to use a mechanical or pharmacological agent depends on Bishop score, parity, contraindications to one of the methods and patient-doctor preference.

Recently, more data are available regarding induction with oral misoprostol (OM) and this method is becoming more popular because OM is effective, safe, convenient, cheap and easy to administer.

If mechanical induction is preferable, either single or double balloon device (DBD) can be used. These methods have been previously studied and neither found to be superior.

A recent study showed that, insertion of the DBD for 6 hours in nulliparous women, results in shorter time to delivery (26 hours vs. 31.4 hours, p=0.015), similar Bishop score after removal ( 5.74 vs. 5.26, p=0.2) without increasing the rate of cesarean deliveries (19% vs 32%, p=0.135) when compared to insertion of the DBD for 12 hours as instructed by the manufacturer. Several studies have shown that a combination of pharmacological and single balloon device results in higher rates to achieve vaginal delivery when compared to each method separately

The investigators hypothesize that with the combination of DBD for 6 hours and OM we will be able to reduce the rate of cesarean deliveries when compared to each method separately.

To date, there are no studies that compared double balloon device with oral misoprostol used concomitantly.

ELIGIBILITY:
Inclusion Criteria:

* unfavourable cervix (Bishop score ≤ 4),
* indication for induction of labor (medical or obstetrical),
* 37 completed gestational weeks,
* vertex presentation,
* singleton pregnancy
* intact membranes.

Exclusion Criteria:

* previous cesarean delivery
* previous uterine surgery (eg: myomectomy)
* noncephalic presentation
* multiple pregnancy
* pre-eclampsia with severe features
* oligohydramnios (Maximal vertical pocket ≤2)
* estimated fetal weight <10% percentile
* any contraindication to Vaginal delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant population
Enrollment: 250 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
the rate of cesarean delivery | from induction until delivery
  percentage of cesarean delivery from all deliveries

SECONDARY OUTCOMES:
Bishop score difference between groups | after 6 hours and after 24 hours
  cervical change evaluation

OTHER OUTCOMES:
time to delivery | from induction to delivery and from ruptured membranes to delivery
  Mean time to delivery
Use of other ripening methods after "failure" of the allocated method | 24 hours after initiation of the treatment
  if the allocated measure was defined as "failed" after 24 hours, other methods will be used to ripen the cervix.
Rate of achieving active phase of labor (≥ 5 cm cervical dilatation) | within 24 hours of initiation
  how many women had more than 5 cm cervical dilatation
Cesarean delivery indication (non progressive labor or non reassuring fetal heart rate NRFHR) | from initiation until cesarean delivery
  what was the indication for surgery
Maternal morbidity | from initiation until delivery
  advanced tears (3rd and 4th degree) post partum hemorrhage uterine rupture, amnionitis
Patient satisfaction - by questioner | within 5 days from delivery
  question addressing pain (bearable or unbearable, was the treatment comfortable for the women and would she do it again if necessary
tachysystole | from initiation until delivery
  more than 5 contractions in 10 min with or without fetal heart rate changes
Neonatal morbidity: | within 5 days from delivery
  neonatal care unit admission, meconium with\without fetal heart rate changes, Apgar 5' <7 ,
use of oxytocin | within 24 hours
  if it was in use at all (yes\no) and if yes- so for how long (time from initiation until delivery)
use of emergent tocolysis | from induction until delivery
  IV atosiban for tachysystole
how many doses of misoprostol | from induction until delivery
  counting the number of administered doses

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Mc, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, Cahill AG, Guise JM, Rouse DJ. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol. 2014 Mar;210(3):179-93. doi: 10.1016/j.ajog.2014.01.026. PMID 24565430
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Schoen C, Navathe R. Failed induction of labor. Semin Perinatol. 2015 Oct;39(6):483-7. doi: 10.1053/j.semperi.2015.07.013. Epub 2015 Sep 2. PMID 26341068
- [Background] Grobman WA, Bailit J, Lai Y, Reddy UM, Wapner RJ, Varner MW, Thorp JM Jr, Leveno KJ, Caritis SN, Prasad M, Tita ATN, Saade G, Sorokin Y, Rouse DJ, Blackwell SC, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Defining failed induction of labor. Am J Obstet Gynecol. 2018 Jan;218(1):122.e1-122.e8. doi: 10.1016/j.ajog.2017.11.556. Epub 2017 Nov 11. PMID 29138035
- [Background] Penfield CA, Wing DA. Labor Induction Techniques: Which Is the Best? Obstet Gynecol Clin North Am. 2017 Dec;44(4):567-582. doi: 10.1016/j.ogc.2017.08.011. PMID 29078939
- [Background] Weeks AD, Navaratnam K, Alfirevic Z. Simplifying oral misoprostol protocols for the induction of labour. BJOG. 2017 Oct;124(11):1642-1645. doi: 10.1111/1471-0528.14657. Epub 2017 May 15. No abstract available. PMID 28342186
- [Background] Salim R, Schwartz N, Zafran N, Zuarez-Easton S, Garmi G, Romano S. Comparison of single- and double-balloon catheters for labor induction: a systematic review and meta-analysis of randomized controlled trials. J Perinatol. 2018 Mar;38(3):217-225. doi: 10.1038/s41372-017-0005-7. Epub 2017 Dec 4. PMID 29203813
- [Background] Husain S, Husain S, Izhar R. Oral misoprostol alone versus oral misoprostol and Foley's catheter for induction of labor: A randomized controlled trial. J Obstet Gynaecol Res. 2017 Aug;43(8):1270-1277. doi: 10.1111/jog.13354. Epub 2017 May 31. PMID 28561987 (Retraction: PMID 34854176 J Obstet Gynaecol Res. 2021 Dec;47(12):4507)
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264